CLINICAL TRIAL: NCT01715428
Title: Effects of Liraglutide on Cardio-Metabolic Risk Markers
Brief Title: Liraglutide and Cardio-Metabolic Risk Markers
Status: Completed | Type: Observational
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Manfredi Rizzo, Assistant Professor, University of Palermo
Other Study IDs: LIRAGLUTIDE UNIPA
Record Dates: First submitted 2012-10-23; First posted 2012-10-29 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Type-2 Diabetes
Keywords: diabetes, cardiovascular risk
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum and plasma samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Liraglutide: administration of liraglutide at 1.2 mg/daily

SUMMARY:
Incretin-based therapies have shown significant effects beyond those on glucose metabolism. We aim in the present study to evaluate the effects of liraglutide on several cardio-metabolic risk markers.

DETAILED DESCRIPTION:
In details, we will evaluate the effects of liraglutide on carotid-intima media thickness, oxidative stress, ghrelin, heat shock proteins and lipoproteins.

ELIGIBILITY:
Inclusion Criteria:

- patients with a diagnosis of type-2 diabetes

Exclusion Criteria:

- severe hepatic or renal diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult subjects with type-2 diabetes
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
carotid intima-media thickness | every four months for a total period of 2 years
  carotid intima-media thickness will be assessed by doppler ultrasonography

SECONDARY OUTCOMES:
changes in oxidative stress markers | after 2 months of therapy
  Serum LOOH levels were evaluated following the oxidation of Fe2+ to Fe3+ in the presence of xylenol orange at 560 nm. Levels of GSH were measured in serum using a spectrophotometric assay based on the reaction of thiol groups with 2,2-dithio-bis-nitrobenzoic acid, while the production of ROS was assessed using fluorescent probe dihydroethidium staining (Sigma).
changes in plasma ghrelin concentrations and heat-shock proteins | after 2 months of therapy
  plasma ghrelin concentrations and heat shock protein 60 were measured by ELISA
changes in atherogenic lipoproteins | after 2 and after 4 months of therapy
  the full LDL subclass profile (from larger and less atherogenic LDL-1 and LDL-2, to smaller denser LDL-3 to LDL-7) was assessed by gel electrophoresis (Lipoprint, Quantimetrix, USA)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Montalto, MD, Study Director — University of Palermo, Italy
Locations (1):
- University Hospital of Palermo, Palermo, Italy

REFERENCES:
- [Derived] Nikolic D, Patti AM, Giglio RV, Chianetta R, Castellino G, Magan-Fernandez A, Citarrella R, Papanas N, Janez A, Stoian AP, Rizvi AA, Rizzo M. Liraglutide Improved Cardiometabolic Parameters More in Obese than in Non-obese Patients with Type 2 Diabetes: A Real-World 18-Month Prospective Study. Diabetes Ther. 2022 Mar;13(3):453-464. doi: 10.1007/s13300-022-01217-z. Epub 2022 Feb 15. PMID 35167051
- [Derived] Nikolic D, Giglio RV, Rizvi AA, Patti AM, Montalto G, Maranta F, Cianflone D, Stoian AP, Rizzo M. Liraglutide Reduces Carotid Intima-Media Thickness by Reducing Small Dense Low-Density Lipoproteins in a Real-World Setting of Patients with Type 2 Diabetes: A Novel Anti-Atherogenic Effect. Diabetes Ther. 2021 Jan;12(1):261-274. doi: 10.1007/s13300-020-00962-3. Epub 2020 Nov 18. PMID 33210276
- [Derived] Rizzo M, Rizvi AA, Patti AM, Nikolic D, Giglio RV, Castellino G, Li Volti G, Caprio M, Montalto G, Provenzano V, Genovese S, Ceriello A. Liraglutide improves metabolic parameters and carotid intima-media thickness in diabetic patients with the metabolic syndrome: an 18-month prospective study. Cardiovasc Diabetol. 2016 Dec 3;15(1):162. doi: 10.1186/s12933-016-0480-8. PMID 27912784
- [Derived] Rizvi AA, Patti AM, Giglio RV, Nikolic D, Amato A, Al-Busaidi N, Al-Rasadi K, Soresi M, Banach M, Montalto G, Rizzo M. Liraglutide improves carotid intima-media thickness in patients with type 2 diabetes and non-alcoholic fatty liver disease: an 8-month prospective pilot study. Expert Opin Biol Ther. 2015;15(10):1391-7. doi: 10.1517/14712598.2015.1067299. Epub 2015 Jul 20. PMID 26195184
- [Derived] Rizzo M, Abate N, Chandalia M, Rizvi AA, Giglio RV, Nikolic D, Marino Gammazza A, Barbagallo I, Isenovic ER, Banach M, Montalto G, Li Volti G. Liraglutide reduces oxidative stress and restores heme oxygenase-1 and ghrelin levels in patients with type 2 diabetes: a prospective pilot study. J Clin Endocrinol Metab. 2015 Feb;100(2):603-6. doi: 10.1210/jc.2014-2291. Epub 2014 Nov 13. PMID 25393640
- [Derived] Rizzo M, Chandalia M, Patti AM, Di Bartolo V, Rizvi AA, Montalto G, Abate N. Liraglutide decreases carotid intima-media thickness in patients with type 2 diabetes: 8-month prospective pilot study. Cardiovasc Diabetol. 2014 Feb 22;13:49. doi: 10.1186/1475-2840-13-49. PMID 24559258